CLINICAL TRIAL: NCT01457716
Title: Pharmacokinetic Pilot Study on Budesonide/Formoterol Device-metered Dry Powder Inhalers, Budesonide/Formoterol Easyhaler and Symbicort Turbuhaler: A Randomised, Open, Single Centre, Single Dose, Crossover Study in Healthy Subjects
Brief Title: Pharmacokinetic Pilot Study on Budesonide/Formoterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3103007
Record Dates: First submitted 2011-09-28; First posted 2011-10-24 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Healthy volunteer study
MeSH Terms: interventions — Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Budesonide/Formoterol Easyhaler A (Experimental)
  Interventions: Drug: Budesonide; Drug: Formoterol; Device: Easyhaler
- Budesonide/Formoterol Easyhaler B (Experimental)
  Interventions: Drug: Budesonide; Drug: Formoterol; Device: Easyhaler
- Budesonide/Formoterol Easyhaler C (Experimental)
  Interventions: Drug: Budesonide; Drug: Formoterol; Device: Easyhaler
- Budesonide/Formoterol Turbohaler Forte (Active Comparator)
  Interventions: Drug: Budesonide; Drug: Formoterol; Device: Turbohaler Forte

INTERVENTIONS:
Drug: Budesonide — Single inhalation
Drug: Formoterol — Single inhalation
Device: Easyhaler — Inhaler device
  Arms: Budesonide/Formoterol Easyhaler A; Budesonide/Formoterol Easyhaler B; Budesonide/Formoterol Easyhaler C
Device: Turbohaler Forte — Inhaler device
  Arms: Budesonide/Formoterol Turbohaler Forte

SUMMARY:
The aim of the study is to assess and compare the Pharmacokinetic (PK) of Budesonide and Formoterol after administration of 3 different product variants of Budesonide/Formoterol Easyhalers and Symbicort turbuhaler.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, 18-55 years of age.
* Normal weight at least 50 kg.

Exclusion Criteria:

* Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological or psychiatric disease.
* Any condition requiring concomitant treatment (including vitamins and herbal products)or likely to need any concomitant treatment during the study
* Any clinically significant abnormal laboratory value or physical finding that may interfere with the interpretation of test results or cause a health risk for the subject if he/she participates in the study.
* Known hypersensitivity to the active substance(s) or to any of the excipients of the drug.
* Pregnant or lactating females.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cmax of Budesonide and Formoterol | 24 hours
AUCt of Budesonide and Formoterol | 24 hours

SECONDARY OUTCOMES:
AUCinf of Budesonide and Formoterol | 24 hours
tmax of Budesonide and Formoterol | 24 hours
t1/2 of Budesonide and Formoterol | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Hietamäki, MSc, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Parexel International GmbH, Berlin, Germany